CLINICAL TRIAL: NCT00272142
Title: Impact of Zinc Supplementation in Low Birth Weight Infants on Severe Morbidity, Mortality and Zinc Status: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: World Health Organization (Other); Linda and Kenneth Pollin Foundation, Inc. (Other)
Responsible Party: Nita Bhandari, Society for Applied Studies
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HNI 04002; C6.181.488
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Diarrhea; Respiratory Infection; Low Birth Weight
Keywords: mortality; hospitalization; diarrhea; respiratory infection; low birth weight; morbidity
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Zinc
Drug: Placebo

SUMMARY:
There are currently no interventions available to substantially reduce the incidence of low birth weight (LBW) apart from increasing the age at marriage, maternal iron supplementation and possibly improved energy intakes.

The current view of the medical and public health community in India is that the immediate focus should be on promoting survival and development of low birth weight infants who have nearly a 6 to 7 fold higher mortality during infancy than those with normal birth weight.

Low serum zinc is associated with increased incidence of diarrhea and pneumonia. There is sufficient evidence in under-threes that during acute illness, zinc supplementation (1-2 recommended dietary allowance [RDA]) reduces incidence of all episodes of diarrhea, severe diarrhea and pneumonia. A number of initial published trials also show significant effect of zinc treatment on pneumonia. With the large and consistent effects of zinc supplementation on the incidence and severity of infections, an effect on child mortality is likely.

Available literature suggests the distinct possibility of reduced neonatal and infant mortality in LBWs receiving 1 RDA of zinc daily. A pilot study in India showed a 54% reduction in mortality in LBW infants. These findings were based on a very small sample and therefore considered insufficient to change policy.

A positive impact in the proposed study will provide an important tool for reduction of infant mortality which is currently stagnant and government acceptance for such a program is likely to be very high. We, the researchers at the Society for Applied Studies, believe this study has the potential for decreasing infant mortality from its current level.

DETAILED DESCRIPTION:
A double blind, randomized, placebo controlled trial is being conducted in which the unit of randomization is 14-28 days old infants. Infants in the intervention group receive 1 RDA of elemental zinc compared to placebo in the control group, from the day of enrollment till 12 months of age.

Infants for enrollment are being identified through daily screening of newborns in two hospitals. Eligible infants are visited at home for enrollment when aged 14-28 days. The mother is trained in supplement administration. A total of 2000 infants will be enrolled.

Infants in the intervention group are being administered a dispersible tablet daily containing 1 RDA of elemental zinc (5 mg elemental zinc per day in infants aged 14 days to 6 months and 10 mg per day for infants older than 6 months) daily till 12 months of age. The placebo contains plain glucose but is similar in taste, color and consistency to the zinc tablet. The tablets are packaged in strips containing 15 tablets each.

Monthly supplies of the supplement are given to the caregiver to be kept at home. The supplement is administered by the caregiver (usually the mother) herself and the method of administration is taught at the time of enrollment. At the end of every four weeks the monitor collects the strips for the previous month and records the supplement intake for the previous month by examining the strips and querying the caregiver.

Three monthly morbidity visits are conducted by a field investigator to obtain information on the hospitalizations and their causes in the last 3 months, healthcare provider visits in the last 1 month, illnesses for which these were made and severity of these illnesses, diarrhea and respiratory morbidity in the previous 24 hours, week and month. If the infant has been hospitalized in the last 3 months, a hospitalization form is filled to ascertain the reason for hospitalization. In case of deaths, an interview is conducted with the caregiver and a verbal autopsy form is filled.

Blood specimens for estimation of plasma zinc, copper and ferritin are being obtained in 15% randomly selected children at baseline and at end study.

Weights and lengths are being obtained in a subset of children at birth, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 14 to 28 days born after 37 weeks of gestation and weighing less than or equal to 2.5 kg at birth (<10th percentile of the National Center for Health Statistics [NCHS] median birth weight)
* Either sex
* Resides within 7 km of the hospital

Exclusion Criteria:

* Likely to leave the area of residence within 6 months of enrollment
* Congenital malformations, congenital heart disease, metabolic disorders, renal diseases, etc.
* Non consent for participation
* Illness requiring hospitalization
* Twins
* Preterm

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
all cause hospitalizations in comparison to infants receiving placebo. | November 2004 to August 2007
illnesses requiring visits to healthcare providers. | November 2004 to August 2007

SECONDARY OUTCOMES:
cause specific hospitalizations for diarrhea and acute lower respiratory infections | November 2004 to August 2007
cause specific health care provider visits for illness | November 2004 to August 2007
all cause mortality in the two groups | November 2004 to August 2007
the proportion of stunted or underweight infants at end study | November 2004 to August 2007
plasma zinc in a subgroup | November 2004 to August 2007
prevalence of diarrheal and respiratory morbidity | November 2004 to August 2007

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, PhD, Principal Investigator — Society for Applied Studies
Locations (1):
- Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Taneja S, Bhandari N, Rongsen-Chandola T, Mahalanabis D, Fontaine O, Bhan MK. Effect of zinc supplementation on morbidity and growth in hospital-born, low-birth-weight infants. Am J Clin Nutr. 2009 Aug;90(2):385-91. doi: 10.3945/ajcn.2009.27707. Epub 2009 Jun 24. PMID 19553296